CLINICAL TRIAL: NCT01557608
Title: Characterization of and Treatment for Chemotherapy-Induced Neuropathy
Brief Title: Characterization and Treatment of Chemotherapy Neuropathy
Acronym: CIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: R01CA151692 (NIH)
Record Dates: First submitted 2012-02-28; First posted 2012-03-19 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Chemotherapy-induced Neuropathy
Keywords: cancer; chemotherapy; photon stimulation; neuropathy; pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Photon stimulation (Experimental)
  Interventions: Procedure: Photon stimulation
- Placebo treatment (Placebo Comparator)
  Interventions: Procedure: Placebo treatment

INTERVENTIONS:
Procedure: Photon stimulation — The LED diode wavelength chosen for this study is 870 nanometers. When activated, the photon stimulator is preset to deliver 1800 Joules in a 7 minute treatment period. Patients will receive a total of 8 treatments, to both feet simultaneously, within a 14 day period depending on their schedule.
  Arms: Photon stimulation
Procedure: Placebo treatment — For patients who receive the placebo treatment, the electronic control unit will be deactivated (i.e., no energy is delivered) even though the indicator lights will be illuminated when the power switch is turned to the "ON" position. Using this procedure, the research nurse who administers the treatments and collects the outcome data will be blinded to the patients' group assignment.
  Arms: Placebo treatment

SUMMARY:
Numbness, tingling, and pain in the hands and feet following the administration of chemotherapy (also called chemotherapy-induced neuropathy (CIN)) is a common problem in oncology patients. However, more information is needed on why patients develop neuropathy and how it impacts their mood, ability to function, and their quality of life. In addition, effective treatments for this problem are not available at the present time. This study will be conducted in two parts. In Part 1, patients who have finished chemotherapy and did or did not develop CIN will be evaluated to determine why some patients do and other patients do not develop CIN. In addition, the impact of CIN on patients' mood, function, and quality of life will be evaluated by comparing patients' reports on these important outcome measures. In addition, genetic markers that contribute to or protect against the development of CIN will be evaluated. Part 2 of this study will test the effects of a new treatment called photon stimulation (also called infrared light therapy) compared to placebo treatment to improve sensations in the feet of oncology patients with CIN. Patients who receive the photon stimulation will have greater improvement in sensation in their feet compared with those who do not receive photon stimulation.

DETAILED DESCRIPTION:
This protocol is designed in two parts. Part 1 will use an "extreme phenotype" approach to evaluate the phenotypic and genotypic characteristics of chemotherapy induced neuropathy(CIN)in a sample of oncology patients who have completed their chemotherapy and did(n=400)and did not (n=200) develop CIN. Patients with and without CIN will be matched, in a 2 to 1 ratio, on their cancer diagnosis and CTX agents administered (i.e., only a platinum compound, only a taxane, or both). Patients will be recruited in cohorts of 30 to 40 to insure that the matching criteria are met and the 2:1 ratio is achieved.

In a single study visit, to take place at the outpatient CTSI CRC (CCRC) at Mt. Zion,participants will be enrolled, complete a battery of sensorimotor tests and questionnaires, and provide a single blood specimen for genomic analysis.

Part 2 will be a pilot study of a randomized, double-blind, placebo-controlled clinical trial (RDBPCT) of photon stimulation in a sample of patients (n=142) with CIN who participated in Part 1. Participants will be randomized to receive the active treatment or the placebo in a series of 8 treatments, lasting 7 minutes each, across a 14-day period. Participants will be assessed at baseline and after the 2nd, 4th, 6th, and 8th treatments with sensory, motor, balance, pain intensity and pain quality measures, mood, and quality of life measures. Blood specimens will be drawn on treatment days 1, 4, 5, and 8 for gene expression.

10.1 * Study design: 10.2 Check

ELIGIBILITY:
Inclusion Criteria:

1. is an adult >18 years of age;
2. has received a platinum compound and/or a taxane;
3. has completed a course of CTX;
4. has changes in sensation and/or pain in their feet of >3 months duration following the completion of CTX;
5. has a rating of >3 on a 0 to 10 numeric rating scale (NRS) on any one of the following sensations from the Pain Qualities Assessment Scale (i.e., numb, tender, shooting, sensitive, electrical, tingling radiating, throbbing, cramping, itchy, unpleasant),91
6. if they have pain associated with the CIN, has an average pain intensity score in their feet of >3 on a 0 to 10 NRS;
7. has a Karnofsky Performance Status (KPS) score of >50;
8. is able to read, write, and understand English; and
9. signs a written informed consent.

Exclusion Criteria:

1. If they have CIN in their hands, because we have no experience treating CIN in patients' hands with photon stimulation and the photon stimulator is designed to provide treatment only to the feet.
2. Women will be excluded if they intend to become or are pregnant or lactating. Men and women will be required to take active measures to prevent pregnancy while on the study.
3. If unwilling to provide the scheduled blood specimens they will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 754 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12-08 (Actual); Study Completion 2015-12-08 (Actual)

PRIMARY OUTCOMES:
Changes over time in light touch sensation | Treatment days 1, 2, 4, 6, and 8
  Light touch sensation will be measured using Semmes Weinstein monofilaments.

SECONDARY OUTCOMES:
Safety measures | Before and after each treatment on days 1 through 8
  Skin will be assessed for redness and swelling.
Changes over time in pain qualities | Treatment days 2, 4, 6, 8
  Pain qualities will be assessed using the Pain Qualities Assessment Scale
Changes over time in average pain intensity | Treatment days 1 through 8
  Average pain will be assessed using a 0 to 10 numeric rating scale.
Changes over time in worst pain intensity | Treatment days 1 through 8
  Worst pain will be assessed using a 0 to 10 numeric rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christine A. Miaskowski, RN, PHD, Principal Investigator — University of California, San Francisco; Bradley Aouizerat, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States